CLINICAL TRIAL: NCT00079391
Title: Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation Followed by T Cell Add-Back for Hematological Malignancies - Effect of Peri-transplant Cyclosporine on Chimerism
Brief Title: Stem Cell Transplantation and T-Cell Add-Back to Treat Bone Marrow Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Minoo Battiwalla, M.D., Staff Clinician, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040112; 04-H-0112 (Other: NIH); NCT00076778 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2014-06

CONDITIONS: Hematologic Malignancies; Bone Marrow Transplant Rejection
Keywords: Chronic Myelogenous Leukemia (CML); Acute Lymphoblastic Leukemia (ALL); Acute Myelogenous Leukemia (AML); Chronic Lymphocytic Leukemia (CLL); Myelodysplastic Syndromes (MDS); Peripheral Blood Stem Cells; Graft-Versus Leukemia/Myeloma; Graft-Versus-Host Disease (GVHD); Cyclosporine; Fludarabine; Leukemia; Myelodysplastic Syndrome; Myeloproliferative Syndrome; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes; Neoplasms, Plasma Cell; Graft vs Host Disease; Leukemia; Lymphoma, Non-Hodgkin | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- allogeneic hematopoietic SCT (Experimental): allogeneic hematopoietic stem cell transplantation (SCT) using Nexell Isolex system
  Interventions: Device: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Device: allogeneic hematopoietic stem cell transplantation — Manipulated Peripheral Blood Stem Cell graft on Day 0. Target CD34+ dose 6 x10e6/kg, (range 3 to 8x10e6/kg) CD3+ dose fixed to 2 x 10e4/kg.
  Other Names: Peripheral Blood Stem Cell Transplant; HSCT; BMT

SUMMARY:
This study will evaluate the safety and effectiveness of stem cell transplantation in which the donor's T cells (a type of lymphocyte, or white blood cell) are removed and then added back. Certain patients with bone marrow malignancies undergo transplantation of donated stem cells to generate new and normally functioning bone marrow. However, T-cells from the donor may see the patient's cells as foreign and mount an immune response to reject them, causing what is called "graft-versus-host-disease" (GVHD). Therefore, in this protocol, T-cells are removed from the donor cells to prevent this complication. However, because T-cells are important in fighting viral infections as well as any remaining malignant cells (called graft-versus-leukemia effect), the donor T-cells are given to the patient (added back) at a later time after the transplant when they can provide needed immunity with less risk of causing GVHD.

Patients between 10 and 55 years of age with acute or chronic leukemia, myelodysplastic syndrome, or myeloproliferative syndrome may be eligible for this study. Prospective participants and their donors are screened with a medical history and physical examination, blood tests (including a test to match for genetic compatibility), breathing tests, chest and sinus x-rays, and tests of heart function. They also undergo a bone marrow biopsy and aspiration. For this procedure, done under local anesthetic, about a tablespoon of bone marrow is withdrawn through a needle inserted into the hipbone.

They undergo apheresis to collect lymphocytes for research studies. This procedure involves collecting blood through a needle in the arm, similar to donating a unit of blood. The lymphocytes are then separated and removed by a cell separator machine, and the rest of the blood is returned through a needle in the other arm.

Before treatment begins, patients have a central intravenous line (flexible plastic tube) placed in a vein in the chest. This line remains in place during the stem cell transplant and recovery period for drawing and transfusing blood, giving medications, and infusing the donated cells. Preparation for the transfusion includes high-dose radiation and chemotherapy. Patients undergo total body irradiation in 8 doses given in two 30-minute sessions a day for 4 days. Eight days before the transplant, they begin taking fludarabine, and 3 days before the procedure they start cyclophosphamide.

DETAILED DESCRIPTION:
Bone marrow stem cell transplant studies carried out by the National Heart Lung & Blood Institute (NHLBI) Bone Marrow Transplantation (BMT) Unit have focused on approaches to optimize the stem cell and lymphocyte dose in order to improve transplant survival and increase the graft-versus-leukemia effect. The aim is to create the transplant conditions that permit rapid donor immune recovery without causing graft-versus-host disease (GVHD) by using reduced post-transplant immunosuppression in conjunction with a transplant depleted of T cells to a fixed low dose, below the threshold known to be associated with GVHD.

We have found that the outcome from transplant is improved by controlling the stem cell (CD34+ cell) and T lymphocyte (CD3+ cell) dose. We use the "Nexell Isolex 300i" system to obtain high CD34+ doses depleted of lymphocytes to a fixed CD3+ T cell dose of 2 x 104/kg. The use of the cell separator and the monoclonal antibodies is covered by an Investigational Device Exemption. A persisting problem with these T cell depleted transplants has been the slow acquisition of full donor T cell engraftment (T cell chimerism). Two previous protocols have failed to increase the speed of donor T cell chimerism. Patients with mixed donor-recipient T cell populations are known to be at higher risk for late graft rejection and leukemic relapse after transplant. Therefore, the achievement of full donor chimerism remains an important therapeutic goal. In this study we will test whether cyclosporine given between day -6 and +21 after transplant can significantly improve day 30 T cell chimerism (the principle end-point). The study also will measure the incidence of acute and chronic GVHD, day 100 transplant related mortality, cytomegalovirus reactivation, relapse, and disease-free survival with appropriate safety stopping rules.

This protocol follows closely previous studies in this series. Three additional modifications will be made however: 1) The first T cell add-back will be delayed until day 60 (instead of day 45) so as to continue to allow a 45 day period without cyclosporine immunosuppression. 2) No day 100 T cell add-back will be given. (In previous studies many patients have, for protocol-defined reasons, not received the second transfusion and there is no evidence that it is required). 3) Patients with high-risk leukemias with a high relapse probability will receive an additional chemotherapy agent prior to transplant using etoposide (VP16) 60mg/kg to improve the chance of remaining in remission.

ELIGIBILITY:
INCLUSION CRITERIA:

RECIPIENT:

* 1. Ages 10-55 years inclusive (but less than 56)
* 2. Chronic myelogenous leukemia (CML) in chronic phase
* 3. Acute lymphoblastic leukemia (ALL) categories

  1. Adults in first remission with high-risk features
  2. All second or subsequent remissions, primary induction failure, partially responding or untreated relapse
* 4. Acute myelogenous leukemia (AML)

  1. AML in first remission Except AML with good risk karyotypes
  2. All AML in second or subsequent remission, primary induction failure and resistant relapse
* 5. Myelodysplastic syndromes categories

  1. refractory anemia with transfusion dependence
  2. refractory anemia with excess of blasts
  3. transformation to acute leukemia, chronic myelomonocytic leukemia
* 6. Myeloproliferative disorders in transformation to acute leukemia
* 7. Chronic lymphocytic leukemia refractory to fludarabine treatment and with bulky progressive disease or with thrombocytopenia (less than or equal to 100,000 /micro L) or anemia (less than or equal to 10g/dl) not due to recent chemotherapy
* 8. Non-Hodgkin's lymphoma including Mantle cell lymphoma relapsing or refractory to current chemotherapy and monoclonal antibody treatment and unsuitable for autologous stem cell transplantation
* 9. No major organ dysfunction precluding transplantation
* 10. Diffusion capacity of lung for carbon monoxide (DLCO) greater than or equal to 60% predicted
* 11. Left ventricular ejection fraction: greater than or equal to 40%
* 12. Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1
* 13. Able to give informed consent
* 14. Negative pregnancy test for women of childbearing age

INCLUSION CRITERIA:

DONOR

* 1. Human leukocyte antigen (HLA) 6/6 identical family donor
* 2. Weight greater than or equal to 18 kg
* 3. Age greater than or equal to 2 or less than or equal to 80 years old
* 4. Fit to receive granulocyte colony -stimulating factor(G-CSF) and give peripheral blood stem cells (normal blood count, normotensive, no history of stroke)

EXCLUSION CRITERIA:

RECIPIENT

* 1. Patient pregnant
* 2. Age less than 10 years and 56 years or more
* 3. Patients with CML in chronic phase who are 41 years or over in whom imatinib mesylate (STI-571)is the treatment of choice
* 4. ECOG performance status of 2 or more
* 5. Severe psychiatric illness
* 6. Major anticipated illness or organ failure incompatible with survival from BMT
* 7. DLCO less than 60% predicted
* 8. Left ventricular ejection fraction: less than 40%
* 9. Serum creatinine greater than 3mg/dl
* 10. Serum bilirubin greater than 4 mg/dl
* 11. HIV positive 12. Debilitation or age making the risk of intensive myeloablative therapy unacceptable

EXCLUSION CRITERIA:

DONOR

* 1. Pregnant or lactating
* 2. Donor unfit to receive G-CSF and undergo apheresis
* 3. HIV positive
* 4. Weight less than 18 kg
* 5. Age less than 2 or greater than 80 years
* 6. Severe psychiatric illness

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minocher Battiwalla, MD, Principal Investigator — NIH National Heart, Lung, and Blood Institute
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Montero A, Savani BN, Shenoy A, Read EJ, Carter CS, Leitman SF, Mielke S, Rezvani K, Childs R, Barrett AJ. T-cell depleted peripheral blood stem cell allotransplantation with T-cell add-back for patients with hematological malignancies: effect of chronic GVHD on outcome. Biol Blood Marrow Transplant. 2006 Dec;12(12):1318-25. doi: 10.1016/j.bbmt.2006.08.034. PMID 17162214
- [Result] Montero A, Savani BN, Kurlander R, Read EJ, Leitman SF, Childs R, Solomon SR, Barrett AJ. Lineage-specific engraftment and outcomes after T-cell-depleted peripheral blood stem cell transplant with Flu/Cy/TBI conditioning. Br J Haematol. 2005 Sep;130(5):733-9. doi: 10.1111/j.1365-2141.2005.05665.x. PMID 16115130
- [Derived] McIver ZA, Yin F, Hughes T, Battiwalla M, Ito S, Koklanaris E, Haggerty J, Hensel NF, Barrett AJ. Second hematopoietic SCT for leukemia relapsing after myeloablative T cell-depleted transplants does not prolong survival. Bone Marrow Transplant. 2013 Sep;48(9):1192-7. doi: 10.1038/bmt.2013.39. Epub 2013 Mar 25. PMID 23524640
- [Derived] McIver Z, Melenhorst JJ, Wu C, Grim A, Ito S, Cho I, Hensel N, Battiwalla M, Barrett AJ. Donor lymphocyte count and thymic activity predict lymphocyte recovery and outcomes after matched-sibling hematopoietic stem cell transplant. Haematologica. 2013 Mar;98(3):346-52. doi: 10.3324/haematol.2012.072991. Epub 2012 Oct 12. PMID 23065508
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2004-H-0112.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow Transplantation Using "Nexell Isolex 300i": Bone marrow stem cell transplant program to improve the outcome of allogeneic Bone Marrow Transplant for hematologic malignancies. Immunosuppression including cyclosporine will be given six days prior to transplant up to 21 days post transplant. cluster of differentiation 34 (CD34) selection and T cell depletion using Isolex 300i immuno-magnetic cell selection and immunosuppression during peri- transplant.
Period: Overall Study
Arm/Group | Bone Marrow Transplantation Using "Nexell Isolex 300i"
Started | 50 (1 of these withdrew after consent.)
Completed | 49
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Bone Marrow Transplantation Using Nexell Isolex 300i: Bone marrow stem cell transplant program to improve the outcome of allogeneic Bone Marrow Transplant for hematologic malignancies. Immunosuppression including cyclosporine will be given six days prior to transplant up to 21 days post transplant. CD34 selection and T cell depletion using Isolex 300i immuno-magnetic cell selection and immunosuppression during peri- transplant.
Arm/Group | Bone Marrow Transplantation Using Nexell Isolex 300i
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Develop Full Donor T Cell Chimerism at Day 30
Description: The proportion of patients who develop full donor CD3+ lymphocyte chimerism by day 30.
  Full chimerism is defined as >95% donor alleles by molecular profiling (Short Tandem Repeat analysis).
Time Frame: Day 30
Population: Per protocol; only patients who survived to day 30 and were evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Bone Marrow Transplantation Using Nexell Isolex 300i
Number analyzed (Participants) | 49
percentage of participants | 44.9

2. Secondary Outcome: Overall Survival
Description: Kaplan Meier estimate of survival
Time Frame: at 5 years post transplant
Measure: Number; unit: percentage of participants
Arm/Group | Bone Marrow Transplantation Using Nexell Isolex 300i
Number analyzed (Participants) | 49
percentage of participants | 47.9

3. Secondary Outcome: Non Relapse Mortality.
Description: Non relapse mortality: death without relapse
  Kaplan Meier estimate
Time Frame: at 5 years post transplant
Measure: Number; unit: percentage of participants
Arm/Group | Bone Marrow Transplantation Using Nexell Isolex 300i
Number analyzed (Participants) | 49
percentage of participants | 21.1

4. Secondary Outcome: Cumulative Incidence of Relapse
Description: Kaplan Meier-estimate of relapse incidence
Time Frame: at 5 years post transplant
Measure: Number; unit: percentage of participants
Groups:
- Bone Marrow Transplantation Using "Nexell Isolex 300i": Bone marrow stem cell transplant program to improve the outcome of allogeneic Bone Marrow Transplant for hematologic malignancies. Immunosuppression including cyclosporine will be given six days prior to transplant up to 21 days post transplant. Cluster of differentiation 34 (CD34) selection and T cell depletion using "Isolex 300i" immuno-magnetic cell selection and immunosuppression during peri- transplant.
Arm/Group | Bone Marrow Transplantation Using "Nexell Isolex 300i"
Number analyzed (Participants) | 49
percentage of participants | 39.8

5. Secondary Outcome: Acute Graft Versus Host Disease (Before Day 60 T Cell Add Back)
Description: Incidence of acute Graft versus host disease (GVHD) grades II-IV (before day 60 T cell add back)
  Modified "Glucksberg" grading
Time Frame: First 60 days
Population: Per protocol
Measure: Number; unit: participants
Groups:
- Bone Marrow Transplantation Using "Nexell Isolex 300i": Bone marrow stem cell transplant program to improve the outcome of allogeneic Bone Marrow Transplant for hematologic malignancies. Immunosuppression including cyclosporine will be given six days prior to transplant up to 21 days post transplant. CD34 selection and T cell depletion using Isolex 300i immuno-magnetic cell selection and immunosuppression during peri- transplant.
Arm/Group | Bone Marrow Transplantation Using "Nexell Isolex 300i"
Number analyzed (Participants) | 49
participants | 20

6. Secondary Outcome: Acute GVHD Overall
Description: Incidence of acute GVHD grades II-IV (before and after T cell add back) Modified Glucksberg grading
Time Frame: First 100 days
Measure: Number; unit: participants
Arm/Group | Bone Marrow Transplantation Using Nexell Isolex 300i
Number analyzed (Participants) | 49
participants | 39

ADVERSE EVENTS:
Time Frame: Overall study
Arm/Group | Bone Marrow Transplantation Using Nexell Isolex 300i
Serious Adverse Events (participants affected / at risk) | 25/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Transplantation Using Nexell Isolex 300i (N=49)
Transplant Related Death (Immune system disorders) | 9 (9)
Hospitalization (Gastrointestinal disorders) | 1 (1)
Hospitalization (Immune system disorders) | 2 (2)
Death (Blood and lymphatic system disorders) | 12 (12)
Life threatening (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Transplantation Using Nexell Isolex 300i (N=49)
Acute GVHD before day 60 (Blood and lymphatic system disorders) | 10 (10)
Chronic GVHD (Blood and lymphatic system disorders) | 22 (22)
Hemorrhagic cystitis (Immune system disorders) | 4 (4)
Cytomegalovirus disease (Immune system disorders) | 37 (37)
Disease Relapse (Blood and lymphatic system disorders) | 18 (18)
Acute GVHD after day 60 (Blood and lymphatic system disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes